CLINICAL TRIAL: NCT01759732
Title: Haploidentical Stem Cell Transplantation With Fixed Dose of T Cells After in Vitro T Cell Depletion Using CD3 Monoclonal Antibody for Children With Acquired Severe Aplastic Anemia
Brief Title: Haploidentical Stem Cell Transplantation for Children With Acquired Severe Aplastic Anemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Ho Joon Im, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMCPHO-SCT1202
Record Dates: First submitted 2012-12-30; First posted 2013-01-03 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2012-12

CONDITIONS: Acquired Aplastic Anemia
Keywords: Aplastic anemia; T cell dose; CD3 depletion; Haploidentical hematopoietic stem cell transplantation
MeSH Terms: conditions — Anemia, Aplastic | interventions — fludarabine; Cyclophosphamide; Antilymphocyte Serum; Filgrastim; Whole-Body Irradiation

ARMS (1):
- HAPLO (Experimental)
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: anti-thymocyte globulin; Biological: filgrastim; Radiation: Total body irradiation; Procedure: CD3-depleted hematopoietic cell transplantation

INTERVENTIONS:
Drug: Fludarabine — 40mg/M2 once daily IV on days -7 to -4
Drug: Cyclophosphamide — 60 mg/kg IV on day-3 and -2
Biological: anti-thymocyte globulin
Biological: filgrastim
  Other Names: Beginning on day 4 and continuing until blood counts recover
Radiation: Total body irradiation — 200 cGy per day on D-5 & -4
Procedure: CD3-depleted hematopoietic cell transplantation — Immunogenetic depletion on CliniMACS

SUMMARY:
Rationale: Fludarabine, cyclophosphamide, anti-thymocyte globulin and low-dose total body irradiation (LD-TBI) may induce the engraftment cross the immunologic barrier in the setting of HLA-haploidentical allogeneic hematopoietic cell transplantation. In addition, depletion of CD3 cells may contribute to prevent developing severe acute graft versus host disease (GVHD) in haploidentical transplantation.

Purpose: Phase II trials to evaluate the efficacy of haploidentical stem cell transplantation with fixed dose of T cells after in vitro T cell depletion using CD3 monoclonal antibody for children with acquired severe aplastic anemia

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of life-threatening marrow failure (severe aplastic anemia) of nonmalignant etiology meeting 2 of the following criteria:

  * Granulocyte count < 500/mm3,
  * Corrected reticulocyte count < 1%,
  * Platelet count < 20,000/mm3
* No HLA-identical family member or closely matched (8 of 8 HLA-locus match) unrelated marrow donor available
* HLA-haploidentical related donor available

Exclusion Criteria:

* Paroxysmal nocturnal hemoglobinuria or Fanconi anemia
* Clonal cytogenetic abnormalities or myelodysplastic syndromes
* Active fungal infections
* HIV positive
* Severe disease other than aplastic anemia that would severely limit the probability of survival during the graft procedure
* Pregnant or nursing

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-09; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
To assess engraftment rate and survival of haploidentical stem cell transplantation with fixed dose of T cells after in vitro T cell depletion using CD3 monoclonal antibody for children with acquired severe aplastic anemia | 2 years posttransplant

SECONDARY OUTCOMES:
To assess engraftment and graft failure | 28 days posttransplant
  Number of patients who failed to engraft by 28 days
To estimate the risk of acute GVHD | 100 days posttransplant
  Number of patients with acute GVHD.
To assess treatment related mortality | 100 days posttransplant
  Number of death after transplantation
To estimate overall survival and failure free survival | 1 year posttransplant

CONTACTS AND LOCATIONS:
Overall Officials: Ho Joon Im, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Burroughs LM, Woolfrey AE, Storer BE, Deeg HJ, Flowers ME, Martin PJ, Carpenter PA, Doney K, Appelbaum FR, Sanders JE, Storb R. Success of allogeneic marrow transplantation for children with severe aplastic anaemia. Br J Haematol. 2012 Jul;158(1):120-8. doi: 10.1111/j.1365-2141.2012.09130.x. Epub 2012 Apr 26. PMID 22533862
- [Background] Tolar J, Deeg HJ, Arai S, Horwitz M, Antin JH, McCarty JM, Adams RH, Ewell M, Leifer ES, Gersten ID, Carter SL, Horowitz MM, Nakamura R, Pulsipher MA, Difronzo NL, Confer DL, Eapen M, Anderlini P. Fludarabine-based conditioning for marrow transplantation from unrelated donors in severe aplastic anemia: early results of a cyclophosphamide dose deescalation study show life-threatening adverse events at predefined cyclophosphamide dose levels. Biol Blood Marrow Transplant. 2012 Jul;18(7):1007-11. doi: 10.1016/j.bbmt.2012.04.014. Epub 2012 Apr 27. PMID 22546497
- [Background] Xu LP, Liu KY, Liu DH, Han W, Chen H, Chen YH, Zhang XH, Wang Y, Wang FR, Wang JZ, Huang XJ. A novel protocol for haploidentical hematopoietic SCT without in vitro T-cell depletion in the treatment of severe acquired aplastic anemia. Bone Marrow Transplant. 2012 Dec;47(12):1507-12. doi: 10.1038/bmt.2012.79. Epub 2012 May 28. PMID 22635243
- [Result] Koh KN, Im HJ, Kim BE, Choi ES, Jang S, Kwon SW, Park CJ, Seo JJ. Haploidentical haematopoietic stem cell transplantation using CD3 or CD3/CD19 depletion and conditioning with fludarabine, cyclophosphamide and antithymocyte globulin for acquired severe aplastic anaemia. Br J Haematol. 2012 Apr;157(1):139-42. doi: 10.1111/j.1365-2141.2011.08924.x. Epub 2011 Nov 5. No abstract available. PMID 22055111
- [Derived] Im HJ, Koh KN, Suh JK, Lee SW, Choi ES, Jang S, Kwon SW, Park CJ, Seo JJ. Refinement of treatment strategies in ex vivo T-cell-depleted haploidentical SCT for pediatric patients. Bone Marrow Transplant. 2015 Feb;50(2):225-31. doi: 10.1038/bmt.2014.232. Epub 2014 Oct 13. PMID 25310303
- See also: Anemia — http://www.nlm.nih.gov/medlineplus/anemia.html
- See also: Fludarabine — http://druginfo.nlm.nih.gov/drugportal/ProxyServlet?mergeData=true&objectHandle=DBMaint&...
- See also: Cyclophosphamide — http://druginfo.nlm.nih.gov/drugportal/ProxyServlet